CLINICAL TRIAL: NCT07097675
Title: The Change in Psychoemotional State of Individuals With Dementia Syndrome Applying Art Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Aušra Sebeikaitė, PhD student, lecturer, Lithuanian University of Health Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-BE10-0004
Record Dates: First submitted 2025-07-09; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Dementia
Keywords: dementia; art therapy; depression; anxiety; stress
MeSH Terms: conditions — Dementia; Depression; Anxiety Disorders | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art Therapy (Experimental)
  Interventions: Behavioral: Art Therapy

INTERVENTIONS:
Behavioral: Art Therapy — Art Therapy Session Plan The sessions are designed to stimulate positive feelings, satisfaction, and calmness while reducing social isolation and fostering group connections. The focus will be on pleasant experiences and positive life moments, with an emphasis on identifying current strengths and capabilities. Every session begins with a sharing activity: "Name three good things that happened this morning" or "Name three things you are grateful for today."
  Session Structure:
  Mood check-in → Warm-up task → Main task → Reflection → Mood check-out.

SUMMARY:
Due to global demographic changes, a notable trend of population aging has emerged, resulting in an increased prevalence of health conditions typically associated with the elderly. One such condition is cognitive impairment-dementia syndrome. Currently, 40,000 cases of dementia are registered in Lithuania (Health Information Centre), with projections estimating 81,000 cases by 2050 [13].

The care of individuals with dementia syndrome requires a holistic approach, incorporating both pharmacological and non-pharmacological interventions. The effectiveness of pharmacological treatment is limited: no highly effective drugs currently exist for Alzheimer's disease (available drugs have limited pathogenetic and symptomatic effects), there are no specific treatments for other forms of dementia, and the long-term use of medications to manage behavioral symptoms is associated with adverse effects. The OECD equates the routine use of neuroleptics with poor quality care [2]. Furthermore, even when medications are prescribed, non-pharmacological interventions should be applied concurrently [5].

One recommended method is arts therapy. Art therapy is a recognized psychosocial treatment that improves attention, perception, memory, and mood in people with dementia. However, there is a lack of studies evaluating the effectiveness of art therapy specifically in improving the psycho-emotional state of individuals with dementia syndrome.

Pharmacological treatments commonly used for dementia syndrome offer limited long-term benefits [23]. As the number of individuals affected by dementia continues to grow, increasing attention is being paid to improving their quality of life, social integration, and emotional well-being through non-pharmacological means. International guidelines recommend creative and artistic activities tailored to individual preferences, skills, and abilities, including music and dance [19]. One of the increasingly recognized interventions is art therapy [5]. Systematic review findings support the inclusion of various psychological interventions in the treatment of individuals with dementia who suffer from depression and/or anxiety disorders [3].

Globally, research most commonly explores the impact of art therapy on cognitive functions, quality of life, behavior, and psychological well-being in individuals with dementia [3; 4]. However, the FEATS scale is rarely used to assess emotional state changes. Although psycho-emotional issues are highly relevant and widely studied, relatively few studies explore these within the context of art therapy. Most existing research is qualitative, with a lack of quantitative studies.

The novelty of this planned study lies not only in the specificity of the participants but also in the application of the FEATS scale. While FEATS is widely used in research, few studies apply this instrument to explore the psycho-emotional state of people with dementia syndrome. The scale's authors and other researchers recommend expanding its use across diverse populations to assess its validity for different patient groups [10; 21].

This study will help reveal the effectiveness of art therapy as a non-invasive and non-pharmacological intervention for improving the psycho-emotional state of individuals with dementia syndrome. The research findings will contribute positively to patient well-being and the advancement of nursing science. Art therapy sessions are expected to improve participants' emotional state and reduce signs of anxiety, depression, and stress. This will provide scientific evidence of the effectiveness of art therapy and allow for the validation of the FEATS scale for assessing the psycho-emotional state of people with dementia syndrome.

DETAILED DESCRIPTION:
Research Aim To determine changes in the psycho-emotional state of individuals with dementia syndrome through the application of art therapy.

Research Objectives

1. To assess the levels of anxiety, depression, and stress in individuals with dementia syndrome before and after art therapy.
2. To evaluate changes in the formal elements of drawings made by individuals with dementia syndrome before and after art therapy.
3. To analyze the relationships between changes in anxiety, depression, and stress levels and changes in the formal elements of drawings among individuals with dementia syndrome.
4. To assess factors potentially associated with changes in anxiety, depression, and stress levels in individuals with dementia syndrome.

Instruments

* For participant selection and assessment of cognitive functions: The Mini-Mental State Examination (MMSE); [7].
* To determine levels of depression, anxiety, and stress before and after art therapy sessions: Lithuanian version of the Depression, Anxiety, and Stress Scales (DASS); [11].
* To assess changes in the formal elements of drawings before and after art therapy sessions: Formal Elements Art Therapy Scale (FEATS); [10].

Sample Size and Justification:

71 participants. The sample size was calculated based on 2022 data from the Lithuanian Health Information Centre.

Study Design and Stages

The following data will be collected from medical records:

* Clinical Data: Primary diagnosis, date of dementia diagnosis, comorbidities, MMSE scores.
* Demographic Data: Gender, age, place of residence, education, occupation, marital status, living situation, and social connections.

The interventions used in this study are not listed in the Lithuanian Ministry of Health's Order No. V-1483 of December 31, 2014, which defines biomedical research methods causing minor and temporary adverse effects on participant health.

Planned Duration and Frequency of Visits Groups of 5-6 participants will meet twice a week for seven weeks.

* First Meeting: Completion of DASS-21 scale and drawing titled "Pick an Apple from the Tree."
* Second to Thirteenth Meetings: Twelve 80-minute art therapy sessions aimed at stimulating positive emotions, enhancing satisfaction and relaxation, and establishing connections with group members. Focus will be placed on pleasant experiences and moments in life, as well as discovering current strengths and abilities. Each session will follow this structure: mood check-in, warm-up task, main task, reflection, mood check-out.
* Fourteenth Meeting: Re-completion of the DASS-21 scale and repeating the drawing "Pick an Apple from the Tree."

Selection of Study Participants and Instruments Used To select study participants, the Mini-Mental State Examination (MMSE); [7] will be used-a short, quick, and easy-to-administer tool that quantitatively assesses cognitive functions [7; 16]. This instrument is widely used in clinical practice and scientific research. Its sensitivity ranges from 0.71 to 0.87 and specificity from 0.81 to 0.96 [15; 1].

The MMSE consists of 11 questions and tasks that analyze seven cognitive domains: orientation in time and space, memorization of three words, attention and calculation, recall of three words, language, and ability to follow simple verbal and written commands. The administration takes approximately 5-10 minutes. For each correct answer or correctly completed task, points are awarded. The fewer the points scored, the more severe the cognitive impairment. The maximum score is 30. A score of ≥25 indicates no cognitive impairment, 20-24 indicates mild impairment, 11-19 indicates moderate impairment, and 0-10 indicates severe cognitive impairment [1].

To assess the psycho-emotional state of the participants, two instruments will be used: the DASS-21 and the FEATS scales, each measuring psycho-emotional states through different approaches.

All instruments are valid, freely available, and do not require author permission for use.

To conduct the study, the following data will be collected:

* Clinical and demographic data from participants (e.g., main diagnosis, date of dementia diagnosis, comorbid conditions, MMSE results, gender, age, place of residence, education, profession, marital status, living situation, and social connections). These data will be recorded using a paper protocol.
* DASS-21 results before and after art therapy sessions, via paper questionnaires.
* Drawings based on the theme "Person Picking an Apple from a Tree."
* Visual expression products created by participants during art therapy sessions. All test and scale data will be evaluated strictly according to methodological guidelines. The collected data will undergo statistical analysis.

The study will be conducted at the Nursing Clinic of Kaunas Clinics of Lithuanian University of Helth Sciences and the Kazys Grinius Nursing and Supportive Treatment Hospital. These institutions were chosen due to enough participants from the target group and because the length of stay of dementia patients allows for the implementation of the planned art therapy intervention.

Field Notes During and after the art therapy sessions, field notes will be kept documenting the study process. These notes will include the researcher's observations, thoughts, questions, and any changes in participants' health status.

Withdrawal from the Study Participants may voluntarily withdraw from the study at any time. No written request will be required. Participation will also be suspended if the researcher or medical staff observes any deterioration in the participant's health.

Recruitment Process The researcher will personally invite patients being treated in the departments and will also work with department staff. Additionally, an invitation poster will be displayed in the department, including the researcher's contact number for those interested.

Informed Consent Procedures Patients at the study sites will receive educational information about art therapy and its potential benefits. Those wishing to participate will be asked to sign an informed consent form. Before beginning, patients whose MMSE score is ≥11 (indicating no severe cognitive impairment) and who are not suffering from unstable chronic somatic illnesses will be selected. Participants must speak Lithuanian to engage in therapy reflections. Individuals meeting these criteria will be invited to participate. Each participant will be informed about the study process, session schedule, and duration.

Potential Benefits Art therapy sessions are expected to evoke positive emotions in participants. They may experience satisfaction, relaxation, and opportunities to form bonds with other group members. This is expected to improve their psycho-emotional state and reduce symptoms of depression, anxiety, and stress.

Potential Risks and Inconveniences Participants may perceive filling out sociodemographic questionnaires and attending art therapy sessions as time-consuming. Traveling to the study site may disrupt daily routines. Sharing personal experiences during therapy reflections may also cause emotional discomfort.

Documentation and Evaluation of Adverse Events

An adverse event is defined as:

* Sudden deterioration in a participant's health during a session.
* Significant psychological discomfort.
* Conflict between the participant and the researcher. If a participant's health worsens during a session, staff at the study site will be called for assistance, and the session will be stopped. All adverse events will be documented in field notes, including the date, researcher involved, description, response, and decisions made.

Data Protection and Confidentiality

The collected data include:

* From medical records: clinical (diagnosis, dementia diagnosis date, comorbidities, MMSE results) and demographic (gender, age, residence, education, profession, marital status, living situation, social ties).
* From participants: DASS-21 results before and after therapy, drawings, and all visual art created during sessions.

All data will be pseudonymized using letter and number codes. If necessary, identifiable data will only be accessible to authorized monitors, ethics committees, or supervising institutions. Coded health data will be available only to the main researchers. Paper questionnaires will be assigned four-digit codes, stored in locked cabinets at the study site, and data will be entered into a OneDrive folder provided by the university and analyzed using SPSS. Access will be password-protected and known only to researchers.

Paper forms, DASS-21 data, and drawings will be stored for 10 years post-study for academic or ethical review, retrospective studies, or dispute prevention. Original data will be destroyed following institutional policy.

If needed, data may be shared with authorized persons, ethics committees, or other supervising institutions. Drawings created during therapy will be returned to participants or their relatives upon request.

De-identified data (study results) will be used in scientific publications and conference presentations.

Participants may withdraw consent at any time before the anonymization of their data. Identifiable data linking participants to their codes will be destroyed immediately after the study ends.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with dementia;
* MMSE ≥11 (mild to moderate cognitive impairment);
* stable somatic condition;
* vision and hearing sufficient to assess cognitive function and to administer interventions;
* familiar with the purpose and conduct of the study;
* signed an informed consent form.

Exclusion Criteria:

* MMSE < 11 points (severe cognitive impairment);
* chronic, unstable somatic conditions;
* Inability to comprehend the tasks;
* Lack of knowledge of the Lithuanian language;
* Refusal to take part in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scales (DASS-21) | Baseline and after 6 weeks
  The DASS-21 is intended to evaluate the severity of depression, anxiety, and stress. It consists of 21 statements divided into three subscales. Each subscale contains seven items grouped by similar content. The depression subscale measures dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest/involvement, anhedonia, and inertia. The anxiety subscale assesses autonomic arousal, physiological responses, situational anxiety, and subjectively experienced anxiety. The stress subscale evaluates difficulty relaxing, nervous tension, sudden sadness, irritability, and excessive reactivity or impatience. The reliability of the Lithuanian version of the DASS-21 is sufficient, making it suitable for use with the Lithuanian population.
  Each item is scored from 0 (no symptom) to 3 (very strong expression of the symptom). Subscale scores are calculated by summing the scores of the respective items.

SECONDARY OUTCOMES:
Formal Elements Art Therapy Scale (FEATS) | Baseline and after 6 weeks
  The FEATS scale evaluates the formal elements of two-dimensional artwork (drawing and painting). It is based on the drawing "Person Picking an Apple from a Tree." Fourteen variables are assessed: color prominence, color fit, energy, space, integration of objects, logic, realism, problem-solving, developmental level, detail of objects and environment, line quality, human figure, position, rotation, and unconscious repetitive motion. Each variable is rated on a Likert scale from 0 to 5. Evaluation is based on structure rather than content, and the FEATS manual outlines specific criteria for each variable.
  Each drawing variable is linked to clinical symptoms, supported by three sources:
  * DSM symptoms that may have graphical correlates in drawings.
  * Literature in art therapy and psychology analyzing spontaneous and directive drawings.
  * Clinical observations of adult psychiatric patients' "Person Picking an Apple from a Tree" drawings.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Norkiene I, Jovarauskaite L, Kvedaraite M, Uppal E, Phull MK, Chander H, Halford K, Kazlauskas E. 'Should I Stay, or Should I Go?' Psychological Distress Predicts Career Change Ideation among Intensive Care Staff in Lithuania and the UK Amid COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Mar 6;18(5):2660. doi: 10.3390/ijerph18052660. PMID 33800903
- [Background] 1. Bikulčius, R. (2014). Application of scales and tests in assessing the physical, mental, and functional condition of the elderly. Gerontology, 15(1), 54-63.
- [Background] 2. de Bienassis, K., Llena-Nozal, A., & Klazinga, N. S. (2020). The economics of patient safety Part III: Long-term care: Valuing safety for the long haul.